CLINICAL TRIAL: NCT03677050
Title: Effect of Individualized Patient Education Including Drinking Advice Using an App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: METC 16-4-141
Record Dates: First submitted 2018-09-14; First posted 2018-09-19 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer
Keywords: Bowel preparation; Colonoscopy; Smart phone application; Patient satisfaction
MeSH Terms: conditions — Colorectal Neoplasms; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: colonoscopist accessing BBPS scores will be blinded; investigator will also assess BBPS scores (not blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): patients receiving standard care (verbal and written instructions) before colonoscopy
- Intervention (Experimental): Patients instructed to use a smart phone patient education app in addition standard care
  Interventions: Other: Smart phone patient education application

INTERVENTIONS:
Other: Smart phone patient education application — Smart phone patient education application including a personalized colonoscopy preparation scheme and information about the procedure.
  Arms: Intervention

SUMMARY:
Study evaluating the effect of a personalized smart phone application in addition to standard care on bowel preparation scores, compared to standard care alone.

DETAILED DESCRIPTION:
Picoprep is a low-volume bowel preparation used to optimize visualization of the colonic mucosa during colonoscopy. Patients referred for a colonoscopy will be scheduled for an intake. During this intake patients receive education about Picoprep and will be asked about their health condition (medical history, medication use). Standard a face-to-face education is given by an intake nurse or doctor. The producers of Picoprep, Ferring BV designed an app including a drinking schedule adapted to the timing of the coloscopy, aiming a lag time between intake of the last Picoprep dose and the scopy of 2-4 hours. We hypothesize that the Boston Bowel Preparation Scale and patient satisfaction will be higher in patients receiving standard education plus using the bowel preparation app versus patients receiving single standard education.

ELIGIBILITY:
Inclusion Criteria:

* Patients refered to our clinic for colonoscopy by general practitioner, colorectal cancer screening programme or outpatient clinic
* Use of regular sodium picosulfate bowel preparation scheme
* Possession of an Android or iOS smart phone

Exclusion Criteria:

* Emergency colonoscopy
* Hospitalized patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Score | During colonoscopy
  Boston Bowel Preparation Score (BBPS) is a validated scale for scoring bowel preparation. Each colonic segment (ascending, transverse, descending) is scored on a scale ranging from 0 to 3, in which a higher value means a cleaner bowel segment. The total score is the sum of the three segment scores (total range 0-9).

SECONDARY OUTCOMES:
Patient satisfaction questionnaire | end of preparation procedure
  Patient satisfaction questionnaire. Several questions in our PSQ (patient satisfaction questionnaire) are based on the PSQ-18. We transformed items from the PSQ-18 to bowel preparation education purposes. The PSQ-18 yields separate scores for each of seven different subscales: General Satisfaction; Technical Quality; Interpersonal Manner; Communication; Financial Aspects; Time Spent with Doctor and Accessibility and Convenience (8, 9). Our PSQ contains items for General Satisfaction (items 3 and 6), Technical Quality (items 8 and 9), Communication (items 1 and 2), Time spent on education (item 7) and Convenience (items 4 and 5). Second, general questions are asked to determine if this was the first time patient received bowel preparation education. And last, for the app users we want to know how they rate the use of the app.
Caecal intubation rate | during colonoscopy
  Total time from insertion of the endoscope to intubation of the caecum.
Adenoma detection rate | during colonoscopy
  percentage of patient in each group in which one or more adenoma(s) are detected.

CONTACTS AND LOCATIONS:
Overall Officials: A.A.M. Masclee, Prof. MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Zander QEW, Reumkens A, van de Valk B, Winkens B, Masclee AAM, de Ridder RJJ. Effects of a Personalized Smartphone App on Bowel Preparation Quality: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Aug 19;9(8):e26703. doi: 10.2196/26703. PMID 34420924